CLINICAL TRIAL: NCT00341783
Title: Assessment of Biologic Parameters in Preparation for Future Malaria Vaccine Trials in Doneguebougou, Mali
Brief Title: Assessment of Biologic Parameters in Preparation for Future Malaria Vaccine Trials in Don gu Bougou, Mali
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902248; 02-I-N248
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2005-07

CONDITIONS: Malaria
Keywords: Plasmodium; Falciparum; Screening; Malaria
MeSH Terms: conditions — Malaria

SUMMARY:
There are about 300-500 million cases of malaria worldwide each year, with 2-3 million deaths. Plasmodium falciparum, one of four types of malaria, is responsible for most of these deaths. Because of increasing resistance of this parasite to drugs and of mosquitoes to insecticides, a vaccine would be valuable in the fight against malaria.

Don gu bougou, Mali, is an area of seasonal malaria transmission that is being investigated as a possible suitable site for testing investigational malaria vaccines. The goal of this study is to characterize the population of this site in terms of common hematologic (blood) and biochemistry parameters that may be used to determine eligibility for participation in vaccine trials. The study will also assess the prevalence of preexisting medical conditions that might affect assessments of vaccine safety and efficacy. Also, the natural immunity to antigens in the investigational malaria vaccines will be determined.

Don gu bougou, Mali, was chosen because of its high malaria rates. Data will be collected at four time-points. At least 50 individuals will be recruited from each of the following age groups: 6 months-5 years; 6-10 years; 11-15 years; and 16-45 years. Village-wide consent will be obtained and about 25 of the 111 family compounds will be randomly selected. Individual consent will also be obtained.

Enrolled volunteers will undergo a baseline medical history and physical examination. Blood will be collected for various tests, and, for women of childbearing age, urine pregnancy tests will be administered.

At each of three followup visits, a brief medical history and physical exam will be conducted. Blood will be drawn for tests. Also, blood, urine, and/or stool tests not done at baseline will be done at one of the followup visits.

DETAILED DESCRIPTION:
Doneguebougou, Mali, is an area of seasonal malaria transmission that is being investigated as a suitable site for testing investigational malaria vaccines. The overall goal of this study is to characterize the population of this site in terms of common hematologic and biochemistry parameters that may be used to determine eligibility for participation in vaccine trials, as well as in terms of preexisting medical conditions and preexisting immunity to potential malaria vaccine antigens, both of which might impact on the assessment of vaccine safety and efficacy. The development of high quality laboratory proficiency to assess these parameters in Mali will also be achieved by this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males or females aged 6 months to 45 years.

Resident of Doneguebougou at the start of the study, and intent to remain a resident for the duration of the study.

Willingness to participate in the study as evidenced by the completed informed consent document.

EXCLUSION CRITERIA:

Clinical evidence of acute life-threatening illness requiring immediate medical care.

Max Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 515
Dates: Start 2002-07; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2002-I-N248.html